CLINICAL TRIAL: NCT03410940
Title: Post-Market Clinical Follow-Up (PMCF) Study of the CLS Brevius Stem With Kinectiv Technology
Brief Title: PMCF Study of the CLS Brevius Stem With Kinectiv Technology
Status: Terminated | Type: Observational
Why Stopped: The production of the device was stopped due to economic reasons. Basic post-market surveillance activities will be continued.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2011-02H
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Femoral Neck Fractures; Prosthesis Failure
Keywords: Total Hip Arthroplasty; CLS Brevius; Kinectiv; Medical Device; Performance; Safety; Hip Prosthesis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Femoral Neck Fractures; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Subjects who received a CLS Brevius Kinectiv stem: Subjects in need of a total hip arthroplasty who met the inclusion/exclusion criteria and received the CLS Brevius Kinectiv stem.
  Interventions: Device: CLS Brevius stem with Kinectiv technology

INTERVENTIONS:
Device: CLS Brevius stem with Kinectiv technology

SUMMARY:
This study is a multi-center, prospective, non-controlled post-market surveillance study. The primary objective of this study is to confirm the safety and performance of the CLS Brevius stem with Kinectiv technology by obtaining implant survivorship and clinical outcomes data for the commercially available stem.

DETAILED DESCRIPTION:
The CLS Brevius Stem with Kinectiv Technology (also referred to as CLS Brevius Kinectiv Stem) is a straight, cementless stem which is based on the successful anchoring philosophy of the CLS Spotorno Stem. In order to be more bone-conserving, the stem was distally shortened by 20% compared to the CLS Spotorno Stem. To restore individual patients' anatomies more accurately, the CLS Brevius Stems are fused with the existing Zimmer Kinectiv Modular Neck Technology.

The objectives of this study are to confirm the safety and performance of the CLS Brevius Kinectiv Stem when used in primary total hip arthroplasty. Safety will be evaluated by monitoring the frequency and incidence of adverse events. Performance will be determined by analyzing the implant survival, overall pain and functional performances, subject quality-of-life and radiographic parameters of study subjects who received the CLS Brevius Kinectiv Stem.

In addition, metal ion levels (titanium and aluminium) will be analyzed pre-operatively and at 6 months, 1, 2 and 5 years in a subset of 70 to 80 patients (30 to 35%).

The primary endpoint is defined as the implant survival at 10 years. Indication: Patients suffering from severe hip pain and disability requiring total hip arthroplasty and who meet the inclusion/exclusion criteria.

Study design: multi-center, prospective, non-controlled. Length of Study: 12 years (20 months enrollment plus 10 years follow-up): follow-up visits at 6 months, 1,2,3,5,7 and 10 years post-operatively.

A maximum total of 230 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age minimum.
* Patient is suffering from severe hip pain and disability requiring primary unilateral or bilateral total hip arthroplasty based on physical exam and medical history.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved 'Informed Consent'.

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient has a total prosthetic hip replacement device (including surface replacement arthroplasty, endoprosthesis etc.) or femoral and/or acetabular osteosynthesis of the affected hip joint(s).
* Patient is: a prisoner, mentally incompetent or unable to understand what participation in the study entails, a known alcoholic or drug abuser, anticipated to be non-compliant
* Acute, chronic local or systemic infections.
* Severe muscular, neural or vascular diseases that endanger the success of the procedure.
* Lack of bony structures proximal or distal to the joint, so that good anchorage of the implant is unlikely or impossible.
* Total or partial absence of the muscular or ligamentous apparatus.
* Any concomitant diseases that can jeopardize the functioning and the success of the implant.
* Allergy to the implanted material, above all to metal (e.g. Vanadium).
* Local bone tumors and/or cysts.
* Pregnancy.
* Skeletal immaturity.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects in need of a total hip arthroplasty, which receive the CLS Brevius Kinectiv stem and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2011-01-07 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Implant survivorship is assessed counting the number of implant revisions | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet
Locations (4):
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna
  - Istituto Ortopedico Galeazzi, Milan
- SPSK im. Prof. A. Grucy, Otwock, Poland
- HUA Santiago, Vitoria-Gasteiz, Spain